CLINICAL TRIAL: NCT01691573
Title: European Pediatric Catheter Ablation Registry
Acronym: EUROPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Principal Investigator, Paolo De Filippo, Principal Investigator, A.O. Ospedale Papa Giovanni XXIII
Other Study IDs: EU01
Record Dates: First submitted 2012-09-11; First posted 2012-09-24 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Cardiac Arrhythmias
Keywords: ablation; procedure; pediatric; european; cardiac; arrhythmias; registry; observational; prospective; catheter; cryoablation; atrioventricular
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of the European Pediatric Catheter Ablation Registry is to collect data on ablation procedures in the European pediatric population in order to improve the management of this subset of patients.

DETAILED DESCRIPTION:
Catheter ablation has revolutionized the management of cardiac arrhythmias in patients and has become first-line therapy for managing many pediatric patients with atrioventricular accessory pathway or atrioventricular nodal-mediated supraventricular tachycardia.

Cardiac ablation in children is not a standardized procedure as in adults as evidence gaps still have to be filled. On a European perspective, lack of a dedicated scientific society has limited so far the collection and sharing of data among the most experienced centers.

Actually there are no sufficient data available about the management of pediatric patients undergoing ablation in clinical practice, in particular regarding indications, methodology and clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients scheduled to any kind of an ablation procedure;
* Patient´s age between 0 and 18 years;
* Legal guardians understand the nature of the procedure, are willing to comply with study follow-up evaluations, and provide written informed consent prior to the procedure.

Exclusion Criteria:

* Patient unable to comply with follow-up schedule;
* Patient has medical conditions that preclude protocol compliance or limit study participation;
* Legal guardian or patient unwilling or unable to provide informed consent.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: European pediatric population
Sampling Method: Probability Sample
Dates: Start 2012-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
To collect data on ablation procedures in the European pediatric population. | After 12 months from the ablation procedure
  Primary outcome will be a combination of efficacy (arrhythmia recurrency) and safety (procedural and late complications)

SECONDARY OUTCOMES:
To describe and compare different ablation methodologies | After 12 months from the ablation procedure
  Rate of index arrhythmia recurrence and rate of complications will be compared for different ablation technology (electroanatomical mapping system vs standard mapping) and for different energy source(radiofrequency vs cryo)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cantù, MD, Principal Investigator — Ospedale Manzoni, Via dell'Eremo 9/11 23900 Lecco, Italy.
Locations (6):
- University Hospital Motol, Prague, Czechia
- Herzzentrum Leipzig GmbH, Leipzig, Germany
- Italy (3):
  - Ospedali Riuniti di Bergamo, Bergamo, BG
  - Ospedali Manzoni, Lecco, LE
  - Ospedale S. Raffaele, Milan, MI
- Leiden University Medical Center, Leiden, Netherlands